CLINICAL TRIAL: NCT05256966
Title: Firefighter Soot, Sauna, and Sweat Excretion Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Minnesota Department of Health (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: A19-131
Record Dates: First submitted 2022-01-28; First posted 2022-02-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Steam Bath; Steam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sauna (Active Comparator): Firefighters/participants based at the station with an existing sauna will be allocated to the intervention arm/sauna group. They will include a sauna session, as per study protocol, which is the intervention.
  Interventions: Other: Sauna (steam)
- Non Sauna (No Intervention): Firefighters/participants based at the stations without a sauna will be allocated to the control arm/Non sauna group. They will not sauna, as per study protocol, as to not receive the study intervention.

INTERVENTIONS:
Other: Sauna (steam) — Steam Sauna
  Arms: Sauna

SUMMARY:
The purpose of the study is to evaluate whether sauna use after active-duty firefighting is effective in reducing exposure to certain harmful chemicals called polycyclic aromatic hydrocarbons (PAHs). PAHs are found in soot and several types are known to be carcinogens.

This study is a cross-sectional pilot study that will be performed in active-duty firefighters. The firefighters will be subdivided into those who will use a sauna immediately after fighting a fire versus those who will not, the latter of which will serve as a metabolism control group. There will thus be two comparison groups within the study: 1) active-duty firefighters using a sauna after fire suppression (sauna group); 2) active-duty firefighters not using a sauna after fire suppression (metabolism control).

DETAILED DESCRIPTION:
Study Rationale

Firefighters are exposed to toxic materials during fire suppression activities and have a higher rate of cancer than the general population, despite a high level of physical fitness. Some studies suggest the use of sauna (infrared or traditional) may increase excretion of harmful and toxic chemicals. Biomonitoring is the measure of chemicals or metabolites present in the human body and is used to evaluate exposure. This proposed study is a biomonitoring pilot study to evaluate the effectiveness of use of a sauna at modulating excretion of select classes of chemicals from firefighters.

One of the most well-established occupational hazards to firefighters is soot, the black particulate matter generated during combustion of organic materials. The chemical composition of soot varies based on the original material undergoing combustion, but the primary organic components of soot comprises a class of compounds known as polycyclic aromatic hydrocarbons (PAHs), which includes many carcinogens.3 PAH exposure can be measured through the analysis of hydroxy metabolites (OH-PAHs) in urine, the methods of which are well-established and have been conducted in the general population and in firefighters in several studies.4-6 The existing literature evaluating excretion of compounds via sweat is suggestive that some compounds may be more quickly eliminated by inducing sweating, such as via use of the sauna. There is a lack of standardization in sweat biomonitoring and further development of these methods is still needed.15 This proposed pilot study will contribute to the biomonitoring literature particularly in the firefighting population by addressing the gaps in knowledge of whether PAHs are excreted in sweat, and whether use of a sauna can affect rates of PAH excretion in firefighters.

Study Objective(s)

Aim 1. This study aims to demonstrate that sauna use immediately after active-duty firefighting will result in measurable (above the level of detection) PAH biomarkers in sweat.

Aim 2. This study secondarily aims to demonstrate that sauna use immediately after active-duty firefighting will result in significantly different mean levels of PAH biomarkers in urine as compared to no use of a sauna.

Study Design

This study is a cross-sectional pilot study that will be performed in active-duty firefighters. The firefighters will be subdivided into those who will use a sauna immediately after fighting a fire versus those who will not, the latter of which will serve as a metabolism control group. There will thus be two comparison groups within the study: 1) active-duty firefighters using a sauna after fire suppression (sauna group); 2) active-duty firefighters not using a sauna after fire suppression (metabolism control).

Subject Population

This study's population is established based on convenience, as the St. Paul Fire Department already has a single station where a sauna has been installed for several decades. The study intervention population will include St. Paul Firefighters working within Station 4, the only station at present where a sauna is installed. The metabolism control group will include St. Paul Firefighters working in stations 7 and 17, who may be called to actively perform at the same fires as the firefighters at Station 4.

St. Paul Firefighters work full-time, on 24-hour shifts, with three different shifts delineated. Station 4 comprises 9 firefighters across 3 shifts, totaling 27 firefighters. The study will be opened to all firefighters in the St. Paul Fire Department, and the Department Chief and department staff will work to schedule individuals enrolled into the study to work at Station 4, 7, or 17.

Inclusion criteria:

1. Willingness to collect urine samples before, during, and/or after work shift
2. Willingness to refrain from eating barbecued or smoked foods during the duration of the study
3. Willingness to use a sauna after active fire suppression and to collect sweat samples at that time

Exclusion criteria:

1. Declined participation in the study
2. Unwilling or do not agree to complete all data collection components of the study
3. Limited from active-duty firefighting (regardless of reason)
4. Medical conditions precluding the use of a sauna
5. Pregnancy (as sauna use is contraindicated in pregnancy)

Number Of Subjects

A minimum of 20 people (10 per group) and a maximum of 60 people (30 per group) will be recruited. As this is a convenience sample, and as not all possible individuals within each sample subpopulation may opt to participate in this study, these samples may be drawn from the same individuals after different active fire runs. Each participant may be asked to provide biosamples up to four times.

The sauna group will comprise 30 urine and 30 sweat samples, whereas the metabolism control group will comprise 30 urine samples, totaling 90 study samples for analysis. The study sample size is limited on resources available for conducting this study and processing samples, and is not intended to meet statistical significance as much as demonstrate differential exposures to PAHs and metabolism of PAHs in the context of this pilot study.

Study Duration

Each subject will be asked to contribute biosamples up to four times. The biosample collection phase is expected to last approximately three months.

The entire study is expected to last 12 months. Study Phases

1. Screening: screening for eligibility and obtaining consent
2. Enrollment: Collection of demographic info and instruction on sample collection
3. Data Collection: Participants collect bio-samples
4. Analysis: MDH analyses of lab samples; statistical analysis to determine study outcomes
5. Results: results provided to participants and analyzed to determine study results
6. Publication: writing and publication of manuscript Statistical And Analytic Plan Statistical testing will comprise a two-tailed t-test (or non-parametric equivalent test if conditions of normality are not met), where statistical significance will be considered at a p-value of <= 0.05.

Aim 1. Detection of PAH parent compounds and metabolites in sweat. Number of detections will be descriptively reported in addition to means and standard deviations of those samples above the report levels.

Aim 2. Comparison of urine PAH biomarkers in sauna group versus metabolism control group. A statistical test of means will be performed on the mean levels of urine PAH biomarkers in the sauna group and the metabolism control group.

The Investigators will use a chi-square test to compare the baseline characteristics of the two groups. If the investigators find a significant difference, the investigators will plan on adjusting for the role of the participant in analysis. Similarly, if the investigators find other baseline characteristic(s) to significantly differ between groups, the investigators will adjust for those variables using multivariate regression that includes treatment group as a variable (Sauna, Metabolism) along with the variables that are unbalanced between the groups.

Statistical analysis will be conducted by the principal investigator (Dr. Zeke McKinney) with the assistance of the Research Methodology Group at the HealthPartners Institute.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to collect urine samples before, during, and/or after work shift
2. Willingness to refrain from eating barbecued or smoked foods during the duration of the study
3. Willingness to use a sauna after active fire suppression and to collect sweat samples at that time

Exclusion Criteria:

1. Declined participation in the study
2. Unwilling or do not agree to complete all data collection components of the study
3. Limited from active-duty firefighting (regardless of reason)
4. Medical conditions precluding the use of a sauna
5. Pregnancy (as sauna use is contraindicated in pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change of PAHs present in sweat | Through study completion, when 90 matched samples have been collected
  This study aims to demonstrate that sauna use immediately after active-duty firefighting will result in a change of PAH biomarkers measurable in sweat.

SECONDARY OUTCOMES:
Change in PAHs present in urine | Through study completion, when 90 matched samples have been collected
  This study secondarily aims to demonstrate that sauna use immediately after active-duty firefighting will result in significantly changed mean levels of PAH biomarkers in urine as compared to no use of a sauna.

CONTACTS AND LOCATIONS:
Overall Officials: Zeke McKinney, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No